# PVP-Guided Decongestive Therapy in HF 2 (PERIPHERAL-HF2)

NCT06495892

July 21st, 2021

### Informed Consent form for patient.

This Informed Consent Form is for the patients who attend the research entitled *Peripheral Venous Pressure-Guided Decongestive Therapy in Heart Failure 2 (PERIPHERAL-HF2)*Study.

This Informed Consent Form has two parts:

Information Sheet (to share information about the research with you)

Certificate of Consent (for signatures if you agree to take part)

You will be given a copy of the full Informed Consent Form

| PART I: Information Sheet Introductio | PART | <b>ˈ l:</b> lnˈ | formation : | Sheet | Introd | luctior |
|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|

| l am, |
|---|
| the chief researcher in the project Peripheral Venous Pressure-Guided Decongestive |
| Therapy in Heart Failure 2 (PERIPHERAL-HF2) at |
| We are doing research on venous pressure (the pressure in your collective veins) in heart |
| failure. I am going to give you information and invite you to be part of this research. You do |
| not have to decide today whether or not you will participate in the research. Before you |
| decide, you can talk to anyone you feel comfortable with about the research. |
| There may be some words that you do not understand. Please ask me to stop as we go |
| through the information and I will take time to explain. If you have questions later, you can |

## Purpose of the research

ask them of me, the study doctor or the staff.)

Heart failure is a chronic disease that causes long term disability and high risk of death. The majority of the symptoms of heart failure is due to excessive fluid collection in the body. One

of the most effective therapies in heart failure patients to alleviate troublesome symptoms are diuretics (urine forcers). These drugs force the patient to urinate and removes this excessive water from the body. Unfortunately, many patients are known to be discharged from the hospital without adequate excess fluid removal, due to the inaccuracy of assessment methods that evaluate whether the right amount of fluid is removed from the body or not. This residual excess fluid in the body is the chief determinant of early re-admissions to the hospital. We believe that we can estimate the need for excess fluid removal by a simple pressure measurement form one of your intravenous lines. If we prove that this approach predicts a better outcome in patients with heart failure, current treatment algorithms for heart failure will change in this direction.

#### Type of Research Intervention

This research will use your demographic data, blood tests and a pressure measurement from one of the intravenous lines that is already put into place. No new intervention will be done and no additional drug will be used in this study.

#### Participant selection

We are screening all adults hospitalized with heart failure to participate in the research.

#### **Voluntary Participation**

Your participation in this research is entirely voluntary. It is your choice whether to participate or not. Whether you choose to participate or not, all the services you receive at this clinic will continue and nothing will change.

**Procedures and Protocol** 

The data recorded in the hospital system during your stay in the hospital will be used and no

new test will be done. After a period, your survival ore readmission status will be checked

from national database.

Duration

The research takes place over 1 to 2 years, but your active presence will not be necessary

after your discharge.

Risks

As there is no new intervention in this study, there is no added risk during the data collecting

process. The healthcare workers will be looking after you and the other participants very

carefully irrespective of your decision on giving consent about your data to be used in the

study.

**Benefits** 

There may not be any benefit for you, but your participation is likely to help us find the answer

to the research question.

Reimbursements

Your participation is free. You will not be given any other money or gifts to take part in this

research.

Confidentiality

The information that we collect from this research project will be kept confidential.

Information about you that will be collected during the research will be put away and no one

but the researchers will be able to see it. Any information about you that will be published in

a scientific journal or presented in a scientific meeting will be completely de-identified and

will not have your name on it.

Sharing the Results

The knowledge that we get from doing this research will be shared with you through

community meetings before it is made widely available to the public. Confidential information

will not be shared.

Right to Refuse or Withdraw

You do not have to take part in this research if you do not wish to do so. It is your choice and

all of your rights will still be respected.

Who to Contact

If you have any questions you may ask them now or later, even after the study has started. If

you wish to ask questions later, you may contact to me.

This proposal has been reviewed and approved by local ethical committee, which is a

committee whose task it is to make sure that research participants are protected from harm.

You can ask me any more questions about any part of the research study, if you wish to. Do

you have any questions?

**PART II:** Certificate of Consent

| I have read the fo | regoing into | ormation, or | it has been read to me. I | have had the op | portunity |
|---|---|---|---|---|---|
| to ask questions a | about it an | d any quest | ions that I have asked ha | ave been answe | red to my |
| satisfaction. I cons | sent volunt | arily to parti | cipate as a participant in t | his research. | |
| Name of Participa | nt | | _ | | |
| Signature of Partic | cipant | | | | |
| Date | | Da | y/month/year | | |
| If illiterate | | | | | |
| A literate witness | must sign (i | if possible, th | nis person should be selec | ted by the partic | cipant and |
| should have no c | connection | to the rese | arch team). Participants | who are illitera | te should |
| include their thum | nb-print as | well. | | | |
| I have witnessed t | the accurat | e reading of | the consent form to the | potential partic | pant, and |
| the individual has | had the opp | portunity to | ask questions. I confirm th | at the individua | has given |
| consent freely. | | | | | |
| Print name of witr | ness | | AND | | |
| Signature of witne | ess | | | | |
| Date | | Day/n | nonth/year | | |
| Thumb print of pa | rticipant | | | | |
| Statement | by | the | researcher/person | taking | consent |
| I have accurately r | ead out the | e informatio | n sheet to the potential p | articipant, and t | o the best |
| of my ability mad | le sure tha | t the partici | pant understands that th | ne following will | be done: |
| 1. My clinical and | laboratory | information | will be used. | | |

3. My survival or re-admission status will be checked trough national database.

2. A pressure is measured from my intravenous line that is already placed.

I confirm that the participant was given an opportunity to ask questions about the study, and all the questions asked by the participant have been answered correctly and to the best of my ability. I confirm that the individual has not been coerced into giving consent, and the consent has been given freely and voluntarily.

A copy of this ICF has been provided to the participant.

| Print Name of Researcher/person tal | king the consent |
|--------------------------------------|------------------|
| Signature of Researcher /person taki | ng the consent |
| Date | Day/month/year |